CLINICAL TRIAL: NCT06059534
Title: Clinical Evaluation of the Improvement of Skin Health Parameters After Oral Intake of DracoBelle Nu in Human Volunteers
Brief Title: Evaluation of the Effects of DracoBelle Nu in Skin Health After Oral Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionos Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DracoBelle_2023
Record Dates: First submitted 2023-08-17; First posted 2023-09-28 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
Keywords: DracoBelleTM Nu; Skin; Aging; Oral; Ingestion; Nutraceutical; Wrinkles; Elasticity; Firmness; Barrier effect; Hydration; Density; Dragonhead; Placebo; Roughness; Fatigue; Pigmentation; Randomized; Blinded
MeSH Terms: conditions — Fatigue | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This group will be provided with placebo capsules for comparative purposes.
  Interventions: Dietary Supplement: Dietary supplementation with placebo.
- DracoBelleTM Nu (Experimental): This group will be provided with DracoBelleTM Nu capsules, which will be compared to the placebo group.
  Interventions: Dietary Supplement: Dietary supplementation with DracoBelleTM Nu.

INTERVENTIONS:
Dietary Supplement: Dietary supplementation with placebo. — Volunteers will be provided with the placebo capsules. For each volunteer, different age-associated skin parameters will be measured with specialized equipment before the treatment and 4, 8 and 12 weeks after the first oral intake of the product.
  Arms: Placebo
Dietary Supplement: Dietary supplementation with DracoBelleTM Nu. — Volunteers will be provided with the DracoBelleTM Nu capsules. For each volunteer, different age-associated skin parameters will be measured with specialized equipment before the treatment and 4, 8 and 12 weeks after the first oral intake of the product.
  Arms: DracoBelleTM Nu

SUMMARY:
The goal of this clinical trial is to study the effects of DracoBelleTM Nu in different skin parameters associated with age. Volunteers will be asked to take either placebo of DracoBelleTM Nu capsules once a day by oral intake for a total period of 12 weeks. Several age-associated skin parameters (skin elasticity, firmness, fatigue, wrinkles, roughness, skin density, hydration, pigmentation and barrier effect) will be measured before the treatment and 4, 8 and 12 weeks after the first oral intake. Data of the placebo and DracoBelleTM Nu group will be analyzed to evaluate the effect of the product DracoBelleTM Nu in the selected age-associated skin parameters.

DETAILED DESCRIPTION:
Skin aging refers to the natural process of changes that occur in the skin as individuals get older. It is a complex biological process influenced by both intrinsic (internal) and extrinsic (external) factors. The signs of skin aging include wrinkles, loss of elasticity and firmness, loss of skin density, reduced skin hydration, altered skin barrier effect and alterations in skin pigmentation. Recent studies show that the consumption of nutraceuticals may improve different parameters associated with skin aging. Recently, it has been shown that daily food supplementation with 200 mg of Moldavian dragonhead dry extract (DracoBelleTM Nu) improved the skin hydration, elasticity and increased skin density. In this placebo-controlled study, the investigators aim to investigate the effects of dietary supplementation with DracoBelleTM Nu in different skin parameters associated with age.

The products will be provided in capsules containing placebo or 200 mg of DracoBelleTM Nu. 50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day, preferably in the morning) for 12 weeks. Different parameters will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. The parameters that will be measured are related to the skin health and skin aging and will be determined as follows:

* The skin elasticity, firmness and fatigue will be measured by the Cutometer in the face skin area.
* Wrinkles (area, length, depth and volume) and roughness of the skin will be measured by the technology Bio3D-MS in the crows-feet and cheek areas.
* The skin density will be measured to determine the thickness of the epidermis and dermis by echography analysis with the UltraScan Echograph in the face skin area.
* Skin hydration will be measured with the Corneometer in the face skin area.
* The skin barrier effect will be measured by quantifying the transepidermal water loss with the Tewameter in the cheek.
* The alterations of the skin pigmentation (area and number of dark spots, and contrast of the dark spots compared to the skin) will be measured with the technology Bio3D-MS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers.
* Between 35-60 years old (both included).
* With noticeable wrinkles.
* Subjects with absence of any infectious disease within the 4 weeks previous to the study.
* Informed of the purpose and the protocol of the study and signed a written informed-consent form.

Exclusion Criteria:

* Diagnosis of any diseases such as cardiovascular disease, chronic kidney disease (CKD), gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease.
* Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females (europa.eu).
* Current smoking habit or history of smoking within the past 1 year.
* History of depression, schizophrenia, alcoholism, drug addiction, or mental illness.
* Current or previous intake of contraceptives, female hormones, obesity drugs, absorption inhibitors, antidepressants, or appetite suppressants.
* History of asthma or autoimmune disease Use of oral hormone therapies ie. cortisone or steroids in the 6 months prior to initiation of the study.
* Abnormal liver function or abnormal renal function.
* Blood pressure >140/90 mmHg or hypertension with intake of a diuretic.
* Any condition judged by the investigator to be unsuitable for participation in the study.
* Subjects refrain from the intake of other oral supplements, including antioxidants, dietary supplements, etc.
* Subjects do not alter their mode of contraception 6 weeks prior and during the study.
* Subjects refrain from any intense or invasive cosmetic treatment, alone or by a beautician, such as intense masks, peelings, and other treatments.
* Subjects are free to follow their usual routine of day and night care products.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Skin elasticity will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin elasticity will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin elasticity will be measured in the face skin area with the Cutometer, and the unit of measurement will be arbitrary units.
Skin firmness will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin firmness will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin firmness will be measured in the face skin area with the Cutometer, and the unit of measurement will be arbitrary units.
Skin fatigue will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin fatigue will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin fatigue will be measured in the face skin area with the Cutometer, and the unit of measurement will be arbitrary units.
Wrinkles will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Wrinkles will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Wrinkles will be measured in the crows feet area with the Bio3D-MS, and the unit of measurement will be arbitrary units.
Roughness will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Roughness will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Roughness will be measured in the crows feet area with the Bio3D-MS, and the unit of measurement will be arbitrary units.
Skin density will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin density will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin density will be measured in the face skin area with the UltraScan Echograph, and the unit of measurement will be arbitrary units.
Skin hydration will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin hydration will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin hydration will be measured in the face skin area with the Corneometer, and the unit of measurement will be arbitrary units.
Skin barrier effect will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin barrier effect will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin barrier effect will be measured in the face skin area with the Tewameter, and the unit of measurement will be arbitrary units.
Skin pigmentation will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake. | Skin pigmentation will be measured before treatment (D0) and at week 4, week 8, and week 12 after the first oral intake of the product.
  50 volunteers will ingest the placebo and 50 volunteers will ingest the product DracoBelleTM Nu by oral intake once a day (one capsule a day) for 12 weeks. Skin pigmentation will be measured in the face skin area with the Bio3D-MS, and the unit of measurement will be arbitrary units.

CONTACTS AND LOCATIONS:
Overall Officials: David Pajuelo Gamez, PhD, Principal Investigator — Hospital La Fe
Locations (1):
- Bionos Biotech S.L., Valencia, Spain

IPD SHARING:
Plan to Share IPD: No